CLINICAL TRIAL: NCT04779437
Title: Using Bayesian Sequential Single Case Methodology to Personalize Low-Intensity Psychological Interventions for Depression: Initial Pilot Work
Brief Title: Bayesian Sequential Single Case Methods to Personalize Low-Intensity Psychological Interventions: Initial Pilot Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Simon Blackwell, Postdoctoral Researcher, Ruhr University of Bochum
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 650
Record Dates: First submitted 2021-02-28; First posted 2021-03-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Depression
Keywords: Depression; Anhedonia; Cognitive Bias Modification; Cognitive Control Training; Bayesian sequential analyses; Single case series
MeSH Terms: conditions — Depression; Anhedonia

STUDY DESIGN:
Intervention Model Description: The study is an exploratory single-case series using a within-subject ABC design, with a baseline phase (A) followed by two intervention phases (B) and (C). Participants are randomly assigned to the order in which they complete the two different interventions.
Masking Description: Two active interventions are used, and both participants and researchers are aware of which intervention participants are completing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imagery Cognitive Bias Modification First (Experimental): After completing two weeks of daily QIDS (baseline phase), participants randomly allocated to this arm will complete two weeks of imagery cognitive bias modification followed by two weeks of cognitive control training. Daily QIDS will be completed throughout the intervention phases.
  Interventions: Behavioral: Imagery Cognitive Bias Modification; Behavioral: Cognitive Control Training
- Cognitive Control Training First (Experimental): After completing two weeks of daily QIDS (baseline phase), participants randomly allocated to this arm will complete two weeks of cognitive control training followed by two weeks of imagery cognitive bias modification. Daily QIDS will be completed throughout the intervention phases.
  Interventions: Behavioral: Imagery Cognitive Bias Modification; Behavioral: Cognitive Control Training

INTERVENTIONS:
Behavioral: Imagery Cognitive Bias Modification — The imagery cognitive bias modification intervention is derived from that developed via experimental psychopathology research (e.g. Holmes et al., 2009) and adapted for clinical applications in the context of depression (e.g. Blackwell & Holmes, 2010; Blackwell et al., 2015). The intervention is a series of training sessions in which participants listen to training scenarios consisting of descriptions of everyday situations, structured so that they start ambiguously but always end positively. Participants are instructed to imagine themselves in the situations described as the scenarios unfold. The training aims to train a bias to automatically imagine positive resolutions for ambiguous situations encountered in daily life.
  Participants will complete one introductory session of the training with the researcher present (in the outpatient center, or via videoconferencing software), then 8 sessions over two weeks completed from home via the study website.
Behavioral: Cognitive Control Training — The cognitive control training is an adaptive Paced Auditory Serial Addition Task (PASAT), adapted from that applied in previous studies (e.g. Siegle et al., 2007; Hoorelbeke et al., 2015; Blackwell et al., 2018). Participants will complete one introductory session of the training with the researcher present (in the outpatient center, or via videoconferencing software), then 8 sessions over two weeks completed from home via the study website.

SUMMARY:
The study is an initial investigation of the feasibility of applying Bayesian sequential analyses to individual participant single-case data for rapid detection of whether or not the individual is benefitting from a low-intensity computerized cognitive training intervention for depression. Patients waiting for, or in follow-up from, outpatient psychological therapy will complete first a two-week period of daily symptom monitoring, followed by two different two-week cognitive training interventions. Data collected will be used to assess feasibility of a future formal case series using Bayesian sequential analyses to determine switching of interventions, and inform the analysis parameters for such a future study.

ELIGIBILITY:
Inclusion Criteria:

* Patient registered at the Ruhr University of Bochum Outpatient Psychotherapy Center ("Zentrum für Psychotherapie", ZPT) in an appropriate phase of treatment (on waiting list/ in follow-up), or from 26/10/22 having had a first consultation ("Beratungsgespräch")
* Aged 18 years or above
* Owning a technical device (e.g. a laptop, computer) that is compatible with the computerized training
* Scoring ≥ 6 on the QIDS (indicating at least mild levels of depressive symptoms)
* Willing and able to complete all study procedures

Exclusion Criteria:

* Existence of a condition or circumstances that would interfere with completion of the study procedures (e.g. severe visual impairment, neurological problem, acute psychosis, or substance withdrawal symptoms)
* Acute crisis with high levels of suicidal ideations or high levels of self-harm, identified either through therapist's assessment or score >1 on item 12 of the QIDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self Report Daily Version (QIDS-daily) | End of intervention (4 weeks post-baseline)
  The QIDS-daily is an adapted version of the QIDS-SR (Rush et al., 2003), which asks about symptoms over the past day and does not include the weight gain/loss items (as used by Holmes et al., 2016). The QIDS-daily will be completed daily over the entire study period, and we will compare the mean and slope of the daily QIDS over the intervention phase to the mean and slope of the daily QIDS in the previous phase.

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self Report (QIDS) | Baseline, pre-intervention (2 weeks post-baseline), between interventions (4 weeks post-baseline), end of study (6 weeks post-baseline)
  The standard QIDS-SR (Rush et al., 2003) is a measure of depression symptoms asking about symptoms over the past seven days.
Dimensional Anhedonia Rating Scale (DARS) | Baseline, pre-intervention (2 weeks post-baseline), between interventions (4 weeks post-baseline), end of study (6 weeks post-baseline)
  The DARS (Rizvi et al., 2015) is a 17-item self-report measure of different facets of anhedonia (desire, motivation, effort and consummatory pleasure) across different hedonic domains (hobbies/past-times, food/drinks, social activities, and sensory experiences).
Positive and Negative Affect Schedule - Positive subscale (PANAS-P) | Baseline, pre-intervention (2 weeks post-baseline), between interventions (4 weeks post-baseline), end of study (6 weeks post-baseline)
  This 18-item positive subscale comprises the Joviality, Self-Assurance, and Attentiveness subscales of the extended PANAS (PANAS-X; Watson & Clark, 1994), and in the current study asks about experience of positive emotions over the past week.
GAD-7 | Baseline, pre-intervention (2 weeks post-baseline), between interventions (4 weeks post-baseline), end of study (6 weeks post-baseline)
  The GAD-7 (Spitzer et al., 2006) is a brief (7 items) self-report anxiety questionnaire designed as a screener for Generalized Anxiety Disorder in primary care.
Positive Mental Health Scale (PMH) | Baseline, pre-intervention (2 weeks post-baseline), between interventions (4 weeks post-baseline), end of study (6 weeks post-baseline)
  The PMH (Lukat et al., 2016) consists of 9 items designed to assess positive mental health.
Prospective Imagery Test (PIT) | Baseline, end of study (6 weeks post-baseline)
  The PIT (Stöber, 2000) is a measure of the vividness with which participants can imagine positive events in their future. In the current study, two 10-item (5 positive and 5 negative) versions are used, with the order counterbalanced across participants.
Daily Expressions of Psychopathology (DEP) | End of intervention (4 weeks post-baseline)
  From 26/10/22 onwards, the DEP is used in addition to the QIDS as a daily measure (completed after the QIDS each day). Nine questions in total were taken (from Wright & Zimmermann, 2021): three depression items, three anxiety items, and three anhedonia items. Participants are asked to rate each item according to much they applied in the past 24 hours, and using a scale from 0 (did not apply at all) to 6 (Applied very strongly). The DEP will be completed daily over the entire study period, and we will compare the mean and slope of the daily DEP over the intervention phase to the mean and slope of the daily DEP in the previous phase.

OTHER OUTCOMES:
Feedback questionnaires | Between interventions (4 weeks post-baseline), end of study (6 weeks post-baseline)
  Feedback questionnaires will be used at the end of each intervention phase, asking about the intervention just completed. Further feedback about the study as a whole will be collected on study completion.
Negative Effects Questionnaire (NEQ) | Between interventions (4 weeks post-baseline), end of study (6 weeks post-baseline)
  The NEQ (Rozental et al., 2019) asks about potential negative effects of psychological interventions. The short (20-item) version is used, adapted to ask about the cognitive training interventions.
Credibility / Expectancy Questionnaires (CEQ) | Baseline, pre-intervention (2 weeks post-baseline), between interventions (4 weeks post-baseline)
  The CEQ (Devilly & Borkovec, 2000) asks participants' assessment of the credibility of the intervention they are about to receive, and their expectation of improvement in symptoms over the course of the intervention. In this study it will be administered before each phase: prior to baseline phase (about completing daily questionnaires), and prior to each intervention phase, about the imagery CBM and Cognitive Control Training as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Simon E Blackwell, Dr. phil., Principal Investigator — Ruhr-Universität Bochum
Locations (1):
- Zentrum für Psychotherapie [Center for Psychotherapy], Mental Health Research and Treatment Center, Ruhr University of Bochum, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available on publication via a suitable repository such as the Open Science Framework, and will be made available to reviewers at the time of submission (or publicly with a pre-print version of the manuscript). Data made available will be the research data reported in the publication, with the exception of any data that could compromise participant anonymity.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Supporting information will be made available on publication via a suitable repository such as the Open Science Framework, and will be made available to reviewers at the time of submission (or publically with a pre-print version of the manuscript).
URL: https://osf.io/qcwfx/